CLINICAL TRIAL: NCT04255797
Title: Chung Shan Medical University Hospital
Brief Title: Effects of Baby Massage on Parenting Stress and Attachment in Premature
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Chung Shan Medical University Hospital, Assistant professor, Chung Shan Medical University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CS19135
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): The experimental group will perform massage in an incubator. The researchers provide a natural plant-based massage oil for the parents.
  Interventions: Behavioral: baby massage

INTERVENTIONS:
Behavioral: baby massage — The steps are as follows:1. Monitor the physiological indicators before massage, 2. Assist premature babies to lie on prone, take off their clothes and diapers, and then apply the baby's massage oil to the hands of both parents to warm them. 3. In the incubator, slight pressure touch the baby's body with warm palms and fingers.

SUMMARY:
This study is an experimental randomized controlled clinical trial. To explore the effect of infant massage on parental pressure and parent-child attachment of premature infants. The intervention time was from 5 days after birth to discharge from premature infants. Data were collected at five time points in longitudinal, before massage (T0), one week (T1), four weeks (T2), and eight weeks ( T3), 12 weeks (T4). Parents in the experimental group were given massage interventions when visiting premature babies, while parents in the control group visited premature babies as usual and contacted premature babies according to general nursing instructions.

DETAILED DESCRIPTION:
The organ development of premature infants is not yet mature, leading to higher morbidity and mortality. Even with advanced technology, parents and families still need to put more effort into taking care of these premature babies so that they can survive. Empirical evidence indicates that baby massage can help parents reduce stress and establish parent-child relationships, but few studies have been applied to parents of premature babies during hospitalization. Based on this, the purpose of this study is: 1. To explore the effect of infant massage on reducing parental pressure; 2. To compare the gender differences of parental pressure; 3. To explore the effect of infant massage on parent-child attachment; 4. Compare the gender difference of parent-child attachment relationship between parents of premature infants. An experimental randomized controlled clinical trial study design was adopted to collect data at five points in time, namely before massage (T0), one week (T1), four weeks (T2), eight weeks (T3), and 12 weeks (T4 ). Using the parental stress scale and parent-child attachment scale. Parents in the experimental group were given massage interventions when visiting premature babies, while parents in the control group were routinely visiting premature babies. The effects of infant massage on parental pressure and parent-child attachment of premature babies at different time points were discussed, and the differences gender of parental pressure and parent-child attachment were compared. The results can increase the empirical research on baby massage, use the empirical knowledge to arouse the attention of nursing staff to baby massage, improve the quality of family-centered care, and pay attention to the needs of parents of different genders.

ELIGIBILITY:
Inclusion Criteria:

1. Single premature infants with a birth week of 30-37 weeks, weighing 1500-2500 grams;
2. The pediatrician assesses the stability of vital signs;
3. Premature infants without congenital abnormalities (such as congenital heart disease) or central nervous system dysfunction (such as intraventricular hemorrhage, epilepsy, etc.); Parents who meet the conditions for premature infants are the study subjects.

Exclusion Criteria:

1. Parents performing kangaroo care;
2. Parents younger than 20 years of age;
3. Parents with mental illness or substance abuse;
4. Single parent father or mother.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Parenting Stress | Up to 12 weeks
  Parents Stress Index-Short Form is a tool for measuring parental stress in premature babies. There are 36 questions in total. Each question uses the Liker's five-point scoring, with a maximum of 180 points and a minimum of 36. The greater the pressure.
Maternal Attachment | Up to 12 weeks
  Maternal Attachment Inventory consists of 26 questions, each of which uses the Liker's four-point scoring method, with a maximum of 104 points and a minimum of 26 points. The higher the score, the better the relationship between mother and baby.

CONTACTS AND LOCATIONS:
Overall Officials: Lien Jen Hwu, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
uncertain

REFERENCES:
- [Result] Alvarez MJ, Fernandez D, Gomez-Salgado J, Rodriguez-Gonzalez D, Roson M, Lapena S. The effects of massage therapy in hospitalized preterm neonates: A systematic review. Int J Nurs Stud. 2017 Apr;69:119-136. doi: 10.1016/j.ijnurstu.2017.02.009. Epub 2017 Feb 14. PMID 28235686